CLINICAL TRIAL: NCT03015324
Title: Biological Effects of Maintenance Usage of Hydroxychloroquine on PAR-4 Levels in Patients With Resected Solid Tumors
Brief Title: Biological Effects of Agent on PAR-4 Levels With Resected Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Peng Wang, MD PhD (Other)
Responsible Party: Sponsor-Investigator, Peng Wang, MD PhD, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-16-MULTI-17
Record Dates: First submitted 2016-12-13; First posted 2017-01-10 (Estimated); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Hydroxychloroquine (Experimental): Hydroxychloroquine
  Interventions: Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Hydroxychloroquine — Hydroxychloroquine

SUMMARY:
Hydroxychloroquine will be administered on an outpatient basis within 12 weeks after primary surgery followed by adjuvant chemotherapy /or radiation therapy (if needed). Hydroxychloroquine will be administered orally at a dose of 400 mg daily for 90 days. Subjects will receive HCQ every day.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor that is surgically resected
* Have completed all planned adjuvant therapy or are not planned for adjuvant therapy
* Age ≥18 years
* ECOG performance status ≤1 (Karnofsky ≥80%)
* Patients must be able to ingest oral medications (crushing and administering via PEG tube is acceptable)
* Patients must have normal organ and marrow function as defined below:
* absolute neutrophil count ≥1,500/mcL
* platelets ≥100,000/mcL
* total bilirubin Less than 1.5 x ULN
* AST(SGOT)/ALT(SGPT) ≤2.5 × institutional upper limit of normal
* creatinine within normal institutional limits OR creatinine clearance ≥50 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* The effects of hydroxychloroquine on the developing human fetus are unknown. For this reason, and because anti-malarial agents as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and four months after completion of hydroxychloroquine administration.
* Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and four months after completion of hydroxychloroquine administration.
* Ability to understand and the willingness to sign a written informed consent document.
* Approval for hydroxychloroquine treatment by an eye doctor, based on a screening eye exam.

Exclusion Criteria:

* Patients with metastatic cancer and/or cancer that is not amenable to surgery.
* Patients with significant malabsorption as determined by the treating physician.
* Patients who are receiving any other investigational agents.
* Patients with known brain metastases are excluded from this clinical trial because of their poor prognosis and because they often develop progressive neurologic dysfunction that would confound the evaluation of neurologic and other adverse events. Patients with primary brain tumors amenable to surgery are allowed on this protocol.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to hydroxychloroquine or received HCQ in the past six months.
* Caution should be taken with the use of hydroxychloroquine and any drugs known to interact with it (Appendix B). Because the lists of these agents are constantly changing, it is important to regularly consult a frequently updated list such as http://medicine.iupui.edu/clinpharm/ddis/table.aspx
* Patients with uncontrolled intercurrent illnesses including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women are excluded from this study.
* HIV-positive patients on combination antiretroviral therapy are ineligible
* Patients that are on enzyme-inducing anti-epileptic medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-08-08 (Actual); Primary Completion 2020-02-03 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
PAR-4 increase | 3 months
  Proportion of patients exhibiting a four-fold increase in PAR-4 levels

SECONDARY OUTCOMES:
Complete Serological Response | 12 months
  Rate of complete serological response in prostate cancer
Progression free survival | 12 months
  Progression free survival in other resected solid tumors

CONTACTS AND LOCATIONS:
Overall Officials: Peng Wang, MD, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky Markey Cancer Center, Lexington, Kentucky, United States